CLINICAL TRIAL: NCT05851001
Title: Effects of Progressive Muscle Relaxation Exercises and Relaxation Music on the Severity of Restless Legs Syndrome and Sleep Quality During Pregnancy: A Randomized Controlled
Brief Title: Effects of Progressive Muscle Relaxation Exercises During Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Esma Yuksel, Research assistant at the Faculty of Health Sciences, Ege University. Midwife, MSc., PhD. (Candidate), Ege University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 16-3-1/13
Record Dates: First submitted 2023-04-27; First posted 2023-05-09 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Restless Legs Syndrome
Keywords: Progressive relaxation exercises; Sleep quality; Relaxation music; Pregnancy
MeSH Terms: conditions — Restless Legs Syndrome; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: Randomized-controlled clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Progressive muscle relaxation (Experimental): A CD recorded by the Turkish Psychological Association was provided to explain relaxation techniques to Progressive muscle relaxation group (PMR ) participants. The CD contains relaxation exercises instructions and there is relaxing music in the background. This CD consists of two parts. The first part(11 minutes) gives short information about the content and how exercises should be done. It consists of information about deep relaxation. In the second part, there are 27 minutes of relaxation exercises accompanied by command with background music.
  PMR exercise consists of four stages: stretching-relaxation (1st stage -approximately 20 minutes), autogenic training - only relaxation (2nd stage approximately 10 minutes), deep breathing training-breathing relaxation (3rd stage approximately 3-4 minutes), rapid relaxation (4th stage--a few seconds).
  Interventions: Other: Progressive Muscle Relaxation exercise
- Relaxation music (Sham Comparator): A CD recorded by the Turkish Psychological Association was provided to RM group participants. It consists of 30 minutes relaxing music only. The participant was asked to just listen to music with without working in a private room.
  Interventions: Other: Muscle relaxation exercise
- Control (No Intervention): In this group, participant were assessed without any other intervention.

INTERVENTIONS:
Other: Progressive Muscle Relaxation exercise — This intervention consists of two parts. The first part (11 minutes) gives short information about the content and how exercises should be done. It consists of information about deep relaxation. In the second part, there are 27 minutes of relaxation exercises accompanied by command with background music.
  Arms: Progressive muscle relaxation
Other: Muscle relaxation exercise — The participant was asked to listen to relaxation music for 30 minutes in a private room.
  Arms: Relaxation music

SUMMARY:
Participants were allocated into three groups; the control group, progressive muscle relaxation (PMR) group and relaxation music (RM) group. The PMR and RM programs were explained toall participants, and the first program was tested under the supervision of the researcher. PMR and RM group participants performed the program daily throughout 4 weeks. Severity of RLS with the International Restless Leg Syndrome Scale (IRLSS) and sleep quality with the Pittsburgh Sleep Quality Index (PSQI) were assessed at baseline, 2 and 4 weeks for all the groups.

DETAILED DESCRIPTION:
A CD recorded by the Turkish Psychological Association was provided to explain relaxation techniques to PMR group participants. The CD contains relaxation exercises instructions and there is relaxing music in the background. This CD consists of two parts. The first part(11 minutes) gives short information about the content and how exercises should be done. It consists of information about deep relaxation. In the second part, there are 27 minutes of relaxation exercises accompanied by command with background music.

PMR exercise consists of four stages: stretching-relaxation (1st stage -approximately 20 minutes), autogenic training - only relaxation (2nd stage approximately 10 minutes), deep breathing training-breathing relaxation (3rd stage approximately 3-4 minutes), rapid relaxation (4th stage--a few seconds). In the first stage, the participant was instructed to first stretch and then relax the specified muscle group (hand, forearm, upper arm, forehead, cheek, nose, chin, neck, chest, shoulder, waist, abdomen, stomach, hip, calf, foot) in sequence. The participant was asked to constantly compare the feeling of tension that shehas just experienced with the feeling of relaxation later.

Another CD recorded by the Turkish Psychological Association was provided to RM group participants. It consists of 30 minutes relaxing music only.The participant was asked to just listen to music with without working in a private room.

ELIGIBILITY:
Inclusion Criteria:

1. diagnosed with RLS by a physician
2. 27 to 34 weeks gestation
3. aged 20 to 35 years
4. able to understand and answer questions in the scale and forms
5. having a CD player

Exclusion Criteria:

* have

  1. vision-hearing problems
  2. chronic disease (hypertension, diabetes mellitus, heart disease, etc.)
  3. any psychiatric diagnosis
  4. multiple pregnancy
  5. rheumatic disease (to avoid difficulties in assessing the severity of RLS)
  6. lumbar hernia and low back pain complaints (to avoid difficulties in assessing the severity of RLS)
  7. varicose veins in the legs (to avoid difficulties in assessing the severity of RLS)

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — We have recruited to study 67 pregnant women.
Enrollment: 67 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2017-04-01 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
Severity of Restless leg syndrome | 10 minutes.
  Severity of Restless leg syndrome was assessed with the International Restless Leg Syndrome Scale Syndrome Scale.

SECONDARY OUTCOMES:
Sleep quality | 24 minutes.
  Sleep quality was examined with the Pittsburgh Sleep Quality Index.

IPD SHARING:
Plan to Share IPD: Undecided
It can be shared upon request.